CLINICAL TRIAL: NCT01023841
Title: Safety and Efficacy of Bimatoprost Solution in Treating Eyelash Loss or Hypotrichosis in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 192024-040
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Results first posted 2013-09-13 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Eyelash Hypotrichosis; Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bimatoprost ophthalmic solution 0.03% (Active Comparator): One drop applied to a sterile single-use-per-eye applicator and applied to upper eyelid margin (where the eyelashes meet the skin) once nightly for 4 months.
  Interventions: Drug: bimatoprost ophthalmic solution 0.03%
- Vehicle Sterile Solution (Placebo Comparator): One drop applied to a sterile single-use-per-eye applicator and applied to upper eyelid margin (where the eyelashes meet the skin) once nightly for 4 months.
  Interventions: Drug: Vehicle Sterile Solution

INTERVENTIONS:
Drug: bimatoprost ophthalmic solution 0.03% — One drop applied to a sterile single-use-per-eye applicator and applied to upper eyelid margin (where the eyelashes meet the skin) once nightly for 4 months.
  Other Names: LATISSE®
  Arms: bimatoprost ophthalmic solution 0.03%
Drug: Vehicle Sterile Solution — One drop applied to a sterile single-use-per-eye applicator and applied to upper eyelid margin (where the eyelashes meet the skin) once nightly for 4 months.
  Arms: Vehicle Sterile Solution

SUMMARY:
This study will evaluate the safety and efficacy of bimatoprost solution 0.03% once daily application to the upper eyelid margins compared with vehicle in treating eyelash loss or hypotrichosis (inadequate or not enough eyelashes) in children.

ELIGIBILITY:
Inclusion Criteria:

* Children who have inadequate eyelashes or have lost their eyelashes as a result of chemotherapy treatment, who completed their chemotherapy (intensive treatment) at least 4 weeks before starting the study, are considered to be at low risk for relapse of their cancer, and are well enough to complete the study
* Children who have minimal to moderate inadequate eyelashes due to alopecia areata
* Adolescents between the ages of 15-17 years who have minimal to marked inadequate eyelashes

Exclusion Criteria:

* Any eye disease or abnormality, eye surgery, permanent eyeliner, eyelash implants.
* Semi-permanent eyelash tint, dye or eyelash extension application within 3 months
* Use of over the counter eyelash growth products within 6 months.
* Use of prescription eyelash growth products (eg, Latisse®)
* Any eye condition that would prevent required ophthalmology exams

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2012-11-02 (Actual); Study Completion 2012-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Newport Beach, California, United States
- São Paulo, Brazil

REFERENCES:
- [Background] Borchert M, Bruce S, Wirta D, Yoelin SG, Lee S, Mao C, VanDenburgh A. An evaluation of the safety and efficacy of bimatoprost for eyelash growth in pediatric subjects. Clin Ophthalmol. 2016 Mar 10;10:419-29. doi: 10.2147/OPTH.S89561. eCollection 2016. PMID 27022239

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost Ophthalmic Solution 0.03% | Vehicle Sterile Solution
Started | 48 | 23
Completed | 47 | 23
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimatoprost Ophthalmic Solution 0.03% | Vehicle Sterile Solution | Total
Number analyzed (Participants) | 48 | 23 | 71
Age, Customized [Number; unit: participants]
  5-11 years | 6 | 3 | 9
  12-17 years | 42 | 20 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 16 | 53
  Male | 11 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event was any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug.
Time Frame: 5 Months
Population: Safety population included all randomized participants who received treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Bimatoprost Ophthalmic Solution 0.03% | Vehicle Sterile Solution
Number analyzed (Participants) | 48 | 23
Percentage of participants | 35.4 | 43.5

2. Secondary Outcome: Change From Baseline Upper Eyelash Length as Measured by Digital Image Analysis (DIA)
Description: Photographs were taken of the eyelashes and assessed using DIA. Length was measured in millimeters (mm). Data from both eyes were averaged for each participant for analysis. A positive change from Baseline indicated longer length (improvement).
Time Frame: Baseline, Month 4
Population: Intent-to-treat population included all randomized participants.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bimatoprost Ophthalmic Solution 0.03% | Vehicle Sterile Solution
Number analyzed (Participants) | 48 | 23
mm
  Baseline | 6.83 (2.568) | 6.04 (2.915)
  Change from Baseline at Month 4 | 1.12 (1.626) | 0.67 (1.846)

3. Secondary Outcome: Change From Baseline in Upper Eyelash Thickness as Measured by DIA
Description: Photographs were taken of the eyelashes and assessed using DIA. Eyelash thickness (fullness) was assessed across both eyes as an average and is measured in millimeters squared (mm^2). A positive change from Baseline indicated fuller eyelashes (improvement).
Time Frame: Baseline, Month 4
Population: Participants from the Intent-to-treat population, that included all randomized participants, with data available at Baseline and Month 4.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Bimatoprost Ophthalmic Solution 0.03% | Vehicle Sterile Solution
Number analyzed (Participants) | 48 | 22
mm^2
  Baseline | 1.20 (0.738) | 1.18 (0.862)
  Change from Baseline at Month 4 | 0.41 (0.535) | 0.05 (0.449)

4. Secondary Outcome: Change From Baseline in Upper Eyelash Darkness as Measured by DIA
Description: Photographs were taken of the eyelashes and assessed using DIA. Eyelash darkness (intensity) was measured in both eyes and averaged for analysis using a scale where 0=black and 255=white. A negative change from Baseline indicated darker eyelashes (improvement).
Time Frame: Baseline, Month 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Intensity units
Arm/Group | Bimatoprost Ophthalmic Solution 0.03% | Vehicle Sterile Solution
Number analyzed (Participants) | 43 | 19
Intensity units
  Baseline | 143.78 (20.446) | 143.44 (25.844)
  Change from Baseline at Month 4 | -15.34 (15.724) | -5.47 (12.289)

5. Primary Outcome: Percentage of Participants With at Least a 1-Grade Improvement From Baseline in the Global Eyebrow Assessment (GEA) Score
Description: The physician evaluated the overall eyelash prominence in both eyes using the GEA 4-point scale: 1= minimal, 2= moderate, 3= marked and 4= very marked. A 1-grade improvement in the GEA score from Baseline indicated improvement.
Time Frame: Baseline, Month 4
Population: Intent-to-treat population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Bimatoprost Ophthalmic Solution 0.03% | Vehicle Sterile Solution
Number analyzed (Participants) | 48 | 23
Percentage of participants | 70.8 | 26.1

ADVERSE EVENTS:
Arm/Group | Bimatoprost Ophthalmic Solution 0.03% | Vehicle Sterile Solution
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/23
Other Adverse Events (participants affected / at risk) | 0/48 | 1/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Bimatoprost Ophthalmic Solution 0.03% (N=48) | Vehicle Sterile Solution (N=23)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0/37 | 1/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.